CLINICAL TRIAL: NCT02112175
Title: Phase 3B, Randomized Trail of Revlimid® (Lenalidomide) Versus Placebo Maintenance Therapy Following Melphalan Prednisone Velcade (Bortezomib) Induction Therapy In Newly Diagnosed Multiple Myeloma
Brief Title: Lenalidomide vs Placebo Maintenance Therapy Following Melphalan Prednisone Velcade® Induction Therapy in NDMM
Acronym: ARUMM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-026
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Lenalidomide; Revlimid; MPV; Melphalan; Prednisone; Velcade; Placebo
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Treatment Arm A: lenalidomide 10 mg/day orally from Days 1 to 21; given in 28-day cycles for up to disease progression.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide

SUMMARY:
The purpose of this study is to compare the safety and efficacy of Lenalidomide versus Placebo maintenance following melphalan, prednisone and velcade induction therapy in newly diagnosed multiple myeloma.

After the study is unblinded, subjects in treatment Arm A (Len 10 mg) will remain on study therapy at the Investigator's discretion and subjects in treatment Arm B (placebo), will be discontinued from study treatment. Subjects who discontinued from study treatment for any reason will enter the LTFU Phase.

DETAILED DESCRIPTION:
The planned total number of evaluable subjects for PFS was approximately 351 (234 in the lenalidomide treatment arm; 117 in the placebo treatment arm) and the study will be conducted in European countries. However, due to the significant enrollment challenges and the changes in the NDMM treatment practices in subjects who are not eligible for transplant, such as the recent approval of Revlimid in NDMM setting, the DMC recommended to close study enrollment. Study enrollment was closed on 12 October 2015.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

Related to initial diagnosis and prior Melphalan Prednisone Velcade (MPV) induction therapy

1. Previously untreated and symptomatic multiple myeloma.
2. All 3 criteria (Durie, 2003) and at least one of the Creatinine Renal insufficiency Anemia lytic Bone lesions or osteoporosis criteria must be met.
3. Measurable disease by protein electrophoresis analyses.
4. All subjects must be treated with a minimum of 6 and a maximum of 9 cycles of MPV induction regimen, and must have achieved at least Partial Response as best overall response and maintained at Melphalan Prednisone Velcade discontinuation. If a subject achieves Complete Response prior to at least 6 cycles, the subject will be eligible, but a minimum of 6 cycles must be administered otherwise.
5. Subjects must not have received any prior anti-myeloma chemotherapy or any investigational agent except 6-9 cycles of induction therapy with Melphalan Prednisone Velcade.
6. Subjects must have cytogenetic (17 p deletion, and 4;14 translocation), β-2 microglobulin and serum albumin (International Staging System) results from their initial diagnosis available at the time of screening.

   Related to the subject
7. Must understand and voluntarily sign the informed consent document prior to the conduct of any study related assessments/procedures,
8. Age ≥ 65 years: if < 65 years of age, the subject must be non eligible for stem cell transplantation,
9. Eastern Cooperative Oncology Group performance status score ≤ 2,
10. Able to adhere to the study visit schedules and other protocol requirements,
11. Females of Childbearing Potential must:

    1. Have two negative pregnancy tests as verified by the study doctor prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after the end of study therapy. This applies even if the subject practices true abstinence2 from heterosexual contact.
    2. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting Investigational Product, during the study therapy (including dose interruptions), and for 28 days after discontinuation of study therapy.
12. Male Subjects must:

    1. Practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female or childbearing potential while participating in the study, during dose interruptions and for at least 28 days following Investigational Product discontinuation, even if he has undergone a successful vasectomy.
    2. Agree to not donate semen during Investigational Product therapy and for 28 days after end of study therapy.
13. All subjects must:

    1. Have an understanding that the study medication could have a potential teratogenic risk.
    2. Agree to abstain from donating blood while taking Investigational Product therapy and following discontinuation of Investigational Product therapy.
    3. Agree not to share study medication with another person.
    4. All female of childbearing potential and male subjects must be counseled about pregnancy precautions and risks of fetal exposure.

Exclusion Criteria:

* The presence of any of the following will exclude the subject from the study enrollment:

  1. Previous treatment with anti-myeloma therapy other than the required 6-9 cycles of Melphalan Prednisone Velcade induction therapy (does not include local radiotherapy, bisphosphonates, or a single short course of steroid [ie, less than or equal to the equivalent of dexamethasone 40 mg/day for 4 days; such a short course of steroid treatment must not have been given within 14 days of randomization]).
  2. Subjects who didn't achieve Partial Response or better after getting at least 6 cycles of Melphalan Prednisone Velcade and at the end of Melphalan Prednisone Velcade whatever the overall response are not eligible.
  3. Prior therapy with immunomodulating or immunosuppressive agents, or epigenetic or desoxyribonucleic acid modulating agents. Subjects who received investigational agents are also excluded.
  4. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
  5. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
  6. Pregnant or lactating females.
  7. Any of the following laboratory abnormalities:

     Absolute neutrophil count < 1,000/L (1.0 x 10*9/L) Untransfused platelet count < 50,000 cells/L (50 x 10*9/L) Serum glutamic oxaloacetic transaminase/alanine aminotransferase or serum glutamic pyruvic transaminase/alanine aminotransferase > 3.0 x upper limit of normal Serum bilirubin levels > 1.5 x upper limit of normal
  8. Renal insufficiency (creatinine clearance < 30 mL/min by Cockcroft-Gault method) or actual creatinine clearance result, or renal failure requiring hemodialysis or peritoneal dialysis.
  9. Prior history of malignancies including skin cancer, other than multiple myeloma.
  10. Prior history of deep venous thrombosis or pulmonary embolus within 3 years of randomization.
  11. Subjects who are unable or unwilling to undergo anti-thrombotic therapy.
  12. Peripheral neuropathy of > Grade 2 severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0.
  13. Known Human Immunodeficiency Virus positivity or active infectious hepatitis, type A, B, or C.
  14. Primary amyloidosis (immunoglobulin light chain) and myeloma complicated by amyloidosis.
  15. Prior allogeneic or autologous stem cell transplantation.
  16. Significant active cardiac disease within the previous 6 months including:

      New York Heart Association class II-IV congestive heart failure Unstable angina or angina requiring surgical or medical intervention Myocardial infarction
  17. Any condition that confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Approximately 6 years
  Is defined as the time from the date of randomization to the date of death due to any cause.

SECONDARY OUTCOMES:
Safety; Adverse Events (AE) [type, frequency, and severity of AEs, and relationship of AEs to investigational product (IP) SAEs, laboratory abnormalities, hospitalizations, and SPMs | Approximately 6 years
  An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study.

CONTACTS AND LOCATIONS:
Overall Officials: Amine Bensmaine, MD, Study Director — Celgene Corporation
Locations (73):
- Belgium (7):
  - Centre Hospitalier EpiCURA - Clinique Louis Caty de Baudour, Baudour
  - AZ-VUB, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - Universitair Ziehenhuis Antwerpen, Edegem
  - Centre Hospitalier de Jolimont-Lobbes, La Louvière-(Haine St-Paul)
  - AZ Nikolaas, Sint-Niklaas
  - Cliniques Universitaires UCL de Mont-Godine, Yvoir
- France (35):
  - CH Argenteuil Victor DupouyHematologie, Argenteuil
  - Centre Hospitalier de la cote basque, Bayonne
  - Hopital Jean Minjoz Hematologie, Besançon
  - Centre Hospitalier de Blois, Blois
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hopital de Fleyriat, Bourg-en-Bresse
  - Hopital A. MorvanHematologie, Brest
  - CHU de la cote de Nacre, Caen
  - CHRU - Hotel Dieu, Clemont-Ferrand Cedex
  - Chu Estaing, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien - Site Gilles de Corbeil, Corbeil-Essonnes
  - Hopital Henri Mondor, Créteil
  - Centre Hospitalier, Dunkirk
  - CHD Vendee, La Roche-sur-Yon
  - CH Hematologie, Le Chesnay
  - Kremlin Bicetre, Le Kremlin-Bicêtre
  - Centre Jean BernardOnco-Hematologie, Le Mans
  - Centre Hospitalier Medecine interne, Le Mans
  - CHRU Hopital Claude Huriez, Lile Cedax
  - CH - Hôpital Dupuytren, Limoges
  - Centre Hospitalier Regional Metz-Thionville Hopital de Mercy, Metz
  - CHU de Nimes, Nîmes
  - CH La Source Onco-Hèmatologie, Orléans
  - Hopital Saint Louis, Paris
  - Groupe Hospitalier Pitié- Salpétrière, Paris
  - CH Perpignan - Hopital Saint-Jean, Perpignan
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier de la Region d'Annecy, Pringy
  - CHRU Hopital sud Medecine Interne, Rennes
  - Centre Hospitalier Yves Le Foll, Saint-Brieuc
  - Hopital civil, Strasbourg
  - CHRU Hôpital de Hautepierre, Strasbourg
  - Institut Universitaire du Cancer IUCT - Oncopole, Toulouse
  - CHRU Hopital BretonneauOnco-hematologie, Tours
  - CHRU Hôpitaux de Brabois, Vandœuvre-lès-Nancy
- Greece (4):
  - Laiko General Hospital of Athens, Athens
  - Alexandra General Hospital of Athens, Athens
  - University of Patras, Pátrai
  - Theagenio Anticancer Hospital of Thessaloniki, Thessaloniki
- Italy (17):
  - Policlinico Sant'Orsola-Malpighi, Bologna
  - Spedali Civili Brescia, Brescia
  - Ospedale Ferrarotto, Catania
  - Clinica Ematologica, A.O.U. San Martino di Genova, Genova
  - Ematologia ed Immunologia, Azienda Ospedaliera Vito Fazzi di Lecce, Lecce
  - Unità Operativa di Oncoematologia, Ospedale di Matera, Matera
  - U.O. di Ematologia e Trapianto di Midollo Osseo, Milan
  - Istituto Nazionale Per Lo Studio E La Cura Dei Tumori Fondazione Giovanni Pascale, Napoli, Campania
  - Policlinico San Matteo Universita Di Pavia, Pavia
  - Ospedale Civile di Piacenza, Piacenza
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Policlinico Umberto I, Roma
  - Ospedale Sant'Eugenio, Rome
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Dipartimento Medicina ed Oncologia Sperimentale - Divisione Universitaria di Ematologia Azienda Ospe, Torino
  - Ospedale Umberto I, Torrette Di Ancona
  - A.O. Universitaria Fondazione Macchi, Varese
- Spain (10):
  - Hospital Sant Pau, Barcelona
  - Hospital Clinic Provincial de Barcelona, Barcelona
  - Hospital virgen de la Arrixaca, El Palmar (murcia)
  - Hospital Virgenes de las Nieves, Granada
  - Hospital La Princesa, Madrid
  - Hospital Costa del Sol, Marbella
  - Hospital Central de Asturias, Oviedo
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Complejo Hospitalario de Santiago, Santiago de Compostela

REFERENCES:
- [Background] Ailawadhi S, Jacobus S, Sexton R, Stewart AK, Dispenzieri A, Hussein MA, Zonder JA, Crowley J, Hoering A, Barlogie B, Orlowski RZ, Rajkumar SV. Disease and outcome disparities in multiple myeloma: exploring the role of race/ethnicity in the Cooperative Group clinical trials. Blood Cancer J. 2018 Jul 6;8(7):67. doi: 10.1038/s41408-018-0102-7. PMID 29980678
- [Background] Dumontet C, Hulin C, Dimopoulos MA, Belch A, Dispenzieri A, Ludwig H, Rodon P, Van Droogenbroeck J, Qiu L, Cavo M, Van de Velde A, Lahuerta JJ, Allangba O, Lee JH, Boyle E, Perrot A, Moreau P, Manier S, Attal M, Roussel M, Mohty M, Mary JY, Civet A, Costa B, Tinel A, Gaston-Mathe Y, Facon T. A predictive model for risk of early grade >/= 3 infection in patients with multiple myeloma not eligible for transplant: analysis of the FIRST trial. Leukemia. 2018 Jun;32(6):1404-1413. doi: 10.1038/s41375-018-0133-x. Epub 2018 Apr 26. PMID 29784907
- [Background] Jain T, Sonbol MB, Firwana B, Kolla KR, Almader-Douglas D, Palmer J, Fonseca R. High-Dose Chemotherapy with Early Autologous Stem Cell Transplantation Compared to Standard Dose Chemotherapy or Delayed Transplantation in Patients with Newly Diagnosed Multiple Myeloma: A Systematic Review and Meta-Analysis. Biol Blood Marrow Transplant. 2019 Feb;25(2):239-247. doi: 10.1016/j.bbmt.2018.09.021. Epub 2018 Sep 20. PMID 30244101
- [Background] Gambella M, Omede P, Spada S, Muccio VE, Gilestro M, Saraci E, Grammatico S, Larocca A, Conticello C, Bernardini A, Gamberi B, Troia R, Liberati AM, Offidani M, Rocci A, Palumbo A, Cavo M, Sonneveld P, Boccadoro M, Oliva S. Minimal residual disease by flow cytometry and allelic-specific oligonucleotide real-time quantitative polymerase chain reaction in patients with myeloma receiving lenalidomide maintenance: A pooled analysis. Cancer. 2019 Mar 1;125(5):750-760. doi: 10.1002/cncr.31854. Epub 2018 Dec 18. PMID 30561775
- [Background] Pegourie B, Karlin L, Benboubker L, Orsini-Piocelle F, Tiab M, Auger-Quittet S, Rodon P, Royer B, Leleu X, Bareau B, Cliquennois M, Fuzibet JG, Voog E, Belhadj-Merzoug K, Decaux O, Rey P, Slama B, Leyronnas C, Zarnitsky C, Boyle E, Bosson JL, Pernod G; IFM Group. Apixaban for the prevention of thromboembolism in immunomodulatory-treated myeloma patients: Myelaxat, a phase 2 pilot study. Am J Hematol. 2019 Jun;94(6):635-640. doi: 10.1002/ajh.25459. Epub 2019 Apr 1. PMID 30859608